CLINICAL TRIAL: NCT06432621
Title: Sugammadex Versus Neostigmine for Recovery of Respiratory Muscle Strength Measured by Ultrasonography in the Postextubation Period in Laparoscopic Cholecystectomy
Brief Title: Role of Sugammadex and Neostigmine for Recovery From Rocuronium
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed wagih Ezzat deusouky, lecturer of anasthesia,intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: MD201/2023
Record Dates: First submitted 2024-04-19; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): patients who will receive sugammadex for recovery from rocuronium and its effect will be assessed by ultrasound and nerve stimulation.
  Interventions: Procedure: using of sugammadex and neostigmine for reversal from rocuronium and assessment of response using ultrasound and nerve stimulation
- Group N (Experimental): patients who will receive neostigmine for recovery from rocuronium and its effect will be assessed by ultrasound and nerve stimulation.
  Interventions: Procedure: using of sugammadex and neostigmine for reversal from rocuronium and assessment of response using ultrasound and nerve stimulation

INTERVENTIONS:
Procedure: using of sugammadex and neostigmine for reversal from rocuronium and assessment of response using ultrasound and nerve stimulation — patients will be randomly divided into two groups using a computer generated random number chart. Group S will receive sugammadex for reversal of rocuronium, whereas Group N will receive neostigmine for reversal of rocuronium using nerve stimulation and ultrasound to asses recovery of respiratory muscle

SUMMARY:
evaluation the reversal of neuromuscular blocking by sugammadex versus neostigmine through assessing the residual neuromuscular blocking effect by ultrasound imaging of expiratory muscle strength and diaphragmatic excursion.

DETAILED DESCRIPTION:
All patients will be assessed preoperatively by careful history taking (history of allergy to rocuronium, neostigmine, or sugammadex), full medical history taking , ASA classification and surgical history Premedication with 2mg midazolam. Anesthesia will be induced with propofol 1-2 mg /kg and fentanyl 1-2 mic/kg. After calibration of TOF (train of four) rocuronium 0.6 mg/kg will be administered, and tracheal intubation will be performed in the absence of train-of four (TOF) count. Rocuronium 0.15mg/kg and Sevoflurane will be used for maintenance of anesthesia.

At the end of the surgery, patients in group A will receive sugammadex (2 mg/kg) and patients in group B will receive neostigmine (50 μg/kg, maximum 5 mg) combined with atropine (25 μg/kg, maximum 2.5 mg) after TOF counts at least exceeding 1 and extubation will be performed in the operating room when the patient is fully awake and fulfilled clinical criteria for extubation.

Diaphragm excursion (DE), reflecting the expiratory and inspiratory muscle strength, respectively, will be measured via ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiology (ASA) physical status classification I and II

Exclusion Criteria:

* 1. American Society of Anesthesiology (ASA) physical status classification III-V 2. renal impairment 3. Significant liver disease (Child-Pugh B or C class) 4. History of chronic obstructive pulmonary disease 5. Known or suspected neuromuscular disease. 6. Cardiac arrhythmia or use of antiarrhythmic drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
effect of sugammadex and neostigmine on reversal of rocuronium | 4 hours
  complete recovery of skeletal muscle assesed by train of four and diaghragmatic excursion by ultrasuond automatically recorded utilizing the TOF monitoring TFIO and diaphragm excursion (DE), reflecting the expiratory and inspiratory muscle strength, respectively, will be measured via ultrasonography (Sonosite M-Turbo) at 3 predefined time points: before induction (baseline levels), TOFR ≥0.9 (postextubation), and after 30 minutes in the PACU.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Ain Shams University, Cairo, Egypt